CLINICAL TRIAL: NCT07126821
Title: A Vision-Language Foundation Model for Brain Disease Diagnosis From Multimodal Data
Status: Recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Xuan Gong, Associate Consultant, Xiangya Hospital of Central South University
Other Study IDs: 2025030464
Record Dates: First submitted 2025-07-31; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Brain (Nervous System) Cancers; Brain Arterial Disease; Neuro-Degenerative Disease; Brain Tumors; Brain Diseases; Neurological di
Keywords: brain tumors; brain cancers; brain diseases; foundation model; diagnosis; prediction; neurological diseases
MeSH Terms: conditions — Neurologic Manifestations; Neoplasms; Intracranial Arterial Diseases; Brain Neoplasms; Brain Diseases; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Interventions — No Interventions

SUMMARY:
The goal of this observational study is to develop an innovative, comprehensive, and explainable AI vision-language foundation model (VLM) to advance the diagnosis and interpretation of brain diseases using multi-modal data. We will include patient demographics, medical imaging data (such as MRI, CT, and PET scans), histopathological data, genomic data when available, and other necessary laboratory examinations and tests to establish a screening and diagnostic model for brain diseases.

DETAILED DESCRIPTION:
Secondary Objective: To establish a comprehensive diagnostic model with uncertainty quantification and automated report generation that covers all brain diseases based on clinical indicators.

Exploratory Objective: To include MRI scans from large-scale populations for model validation.

ELIGIBILITY:
Inclusion Criteria:

Patients with brain diseases:

* Patients with brain tumors were pathologically diagnosed.
* Patients with other brain diseases were correctly diagnosed.
* The clinical case data of all patients were complete.

Non-brain disease population:

* All patients have complete clinical case data, complete brain MRI, no history brain diseases, no brain surgery or other brain diseases that affect the diagnosis and observation of MR imaging.

Exclusion Criteria:

* Cases in which MRI were incomplete or with significant noise and artifacts.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with brain disease or Non-disease condition
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Brain Disease Diagnostic performance | Perioperative
  This study will evaluate how accurately the AI model can identify and differentiate between: 1. Brain tumors including gliomas, glioneuronal tumors, and neuronal tumor, meningioma, germ cell tumors, embryonal tumors, tumors of the sellar region, pineal region tumors, mesenchymal, non-meningothelial tumors, choroid plexus tumors, hematolymphoid tumors, cranial and paraspinal nerve tumors, melanocytic tumors and brain metastases based on WHO CNS 5 classification; 2. Brain diseases apart from brain tumors such as brain arterial disease, neurodegenerative disorders, etc.; 3. Normal brain findings; The model's performance will be assessed using sensitivity, specificity, F1-score AUC-ROC. Diagnostic ability of AI model will be compared against with pathological diagnosis(if possible), final clinical diagnoses by neurologists or radiologists.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No